CLINICAL TRIAL: NCT01689792
Title: A Multi-centre, Randomised, Investigator-blinded Study Comparing the Polyp Detection Rate of Two Different Types of Bowel Preparation: a 2-litre Solution (MOVIPREP®) Versus a Hyperosmotic and Stimulant Combined Low Volume Bowel Preparation (Sodium Picosulfate and Magnesium Citrate)
Brief Title: A Multi-centre Study Comparing the Polyp Detection Rate of Two Different Types of Bowel Preparation: a 2-litre Solution (MOVIPREP®) Versus a Hyperosmotic and Stimulant Combined Low Volume Bowel Preparation (Sodium Picosulfate and Magnesium Citrate)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NOR-01/2011 (PDR)
Record Dates: First submitted 2012-09-12; First posted 2012-09-21 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CitraFleet (Active Comparator): Administration of CitraFleet
  Interventions: Drug: CitraFleet
- MOVIPREP (Experimental): Administration of MOVIPREP
  Interventions: Drug: MOVIPREP

INTERVENTIONS:
Drug: MOVIPREP
  Arms: MOVIPREP
Drug: CitraFleet
  Arms: CitraFleet

SUMMARY:
To compare the polyp and adenoma detection rate of MOVIPREP versus an oral Sodium Picosulfate/Magnesium Citrate solution.

ELIGIBILITY:
Inclusion Criteria:

* Patient's written informed consent must be obtained prior to inclusion.
* Male or female outpatients or inpatients aged 40 to 80 years with an indication for complete colonoscopy.
* Willing to undergo a colonoscopy for diagnostic or surveillance purposes
* Patients with a known personal of familial risk of colon neoplasia, willing to undergo a screening colonoscopy
* Willing, able and competent to complete the entire procedure and to comply with study instructions.
* Females of childbearing potential must employ an adequate method of contraception.

Exclusion Criteria:

* History of gastric emptying disorders.
* History of ileus, toxic megacolon, gastrointestinal obstruction and colonic perforation.
* History of phenylketonuria.
* Known glucose-6-phosphate dehydrogenase deficiency.
* Known hypersensitivity to macrogol 3350, sodium sulphate or ascorbic acid/sodium ascorbate.
* History of colonic resection.
* Requirement for permanent medication and associated stable serum concentrations (e.g. neuroleptic drugs).
* Presence of congestive heart failure (NYHA III + IV).
* Acute life-threatening cardiovascular disease.
* Documented history of severe renal insufficiency (creatinine clearance <30 ml/min).
* Other contraindication described in the summary of product characteristics (SmPC) of either preparation.
* Patient has a condition, clinically significant laboratory results, or is in a situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly.
* Application of any unlicensed medication within the previous 3 months or participation in any other research study in the last 3 months.
* Females who are pregnant, nursing or planning a pregnancy.
* Patients who, in the opinion of the investigator, may not be compliant with the study requirements.
* Previous participation in this clinical study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Polyp detection rate | At colonoscopy
  Polyp detection rate defined as number of patients with at least one polyp or flat lesion as recorded by the endoscopist

SECONDARY OUTCOMES:
Adenoma Detection Rate (ADR) | At the Colonoscopy
  ADR, (including flat lesions) defined as number of patients with at least one adenoma as recorded by the pathologist in relation to the total analysis population
ADR and PDR by location | at the colonoscopy
  ADR and PDR by location:
  * left sided (rectum, colon sigmoideum, colon decendens, left half of colon transversum
  * right-sided (right half of colon transversum, colon ascendens, caecum
Cancer detection rate | at the colonoscopy
  Cancer detection rate, defined as number of patients with at least one malignancy in relation to the total analysis population
Flat lesion only detection rate | at the colonoscopy
  Flat lesion only detection of the patients
Advanced risk lesion detection rate | at the colonoscopy
  Advanced risk lesion detection rate (lesions >1 cm, low grade and/or villous
Colonoscopy completion rate | at the colonoscopy
  The rate of colonoscopy completion
Colon cleansing quality | at the colonoscopy
  Colon cleansing quality as reported by the gastroenterologist, according to the Harefield Cleansing Scale©
Acceptability and tolerability of medication using patient questionnaires | Throughout the study
  The acceptability and tolerability of the study medication taken by the patients throughout the study using specified patient questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Fishbach, MD, Principal Investigator — Klinikum Aschaffenburg-Alzenau
Locations (1):
- Klinikum Aschaffenburg, Aschaffenburg, Germany

REFERENCES:
- [Derived] Pohl J, Halphen M, Kloess HR, Fischbach W. Impact of the quality of bowel cleansing on the efficacy of colonic cancer screening: a prospective, randomized, blinded study. PLoS One. 2015 May 7;10(5):e0126067. doi: 10.1371/journal.pone.0126067. eCollection 2015. PMID 25950434